CLINICAL TRIAL: NCT00408642
Title: An Enhanced Adherence Support Programme for HAART
Brief Title: An Enhanced Adherence Support Programme for Highly Active Antiretroviral Therapy (HAART)
Acronym: eASP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Dr Salim S Abdool Karim, Director, Centre for the AIDS Programme of Research in South Africa
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CAP 058
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: HIV Infections
Keywords: adherence; treatment; antiretroviral; HAART; HIV; Treatment Naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): enhanced adherence support for patients initiating antiretroviral therapy
  Interventions: Behavioral: Enhanced adherence support
- 2 (Active Comparator): standard adherence support
  Interventions: Behavioral: Standard adherence support

INTERVENTIONS:
Behavioral: Enhanced adherence support — The enhanced adherence support intervention consists of 5 one-on-one, Information-Motivation-Behavioral Skills (IMB) theory-based counseling sessions, as well as a problem-solving card which summarizes key messages and strategies. The counseling sessions are given at key points post-initiation of therapy: at baseline, 2 weeks, 2 months, 3 months, and 6 months. Three brief weekly ART planning sessions are conducted post-initiation of therapy.
  Arms: 1
Behavioral: Standard adherence support — The control arm receives the standard of care adherence support which consists of three group counseling adherence sessions conducted prior to initiation of therapy.
  Arms: 2

SUMMARY:
In southern Africa, TB is the most common first AIDS-defining condition. Initiating Antiretroviral therapy (ART) in HIV positive TB patients will lead to the inclusion of the majority of HIV/AIDS patients currently fulfilling the criteria for therapy. Establishing an effective intervention to increase treatment adherence in this group is essential for the successful roll out of ART in the region. This proposed randomized controlled study aims to compare the effectiveness of two adherence support programmes (ASP) for use in patients with HIV-related TB in the context of CAPRISA AIDS Treatment (CAT)programme in KwaZulu-Natal, South Africa; the enhanced adherence support programme (E-ASP) or the standard adherence support programme (S-ASP).

S-ASP consists of three counselor presented, group education sessions. E-ASP is an extension of S-ASP and is based on the Information-Motivation-Behavioral Skills (IMB) Model of Adherence to Antiretroviral Therapy, a theoretical model initially developed to reduce HIV risk behavior. The E-ASP will consist of several interconnected components: 1) development and maintenance of an educational and supportive milieu at the CDC Clinic, 2) provision of five structured educational, support and behavioral skills building sessions, and (3) three weekly ART planning sessions.

DETAILED DESCRIPTION:
Enhanced Adherence Support (E-ASP)

All patients will receive sessions one and two of the Standard ASP. Following randomization, the intervention (experimental) arm patients receive the E-ASP described below and the standard of care (control) arm patients receive session three of the S-ASP.

Two health educators are employed and trained to administer E-ASP. The goal of the E-ASP is to identify and address patient deficits in information, motivation, and behavioural skills that inhibit consistent and correct self-administration of ARV medications, including those skills required to adhere to the clinic visit schedule. By using specific motivational techniques (Motivational Interviewing) and structured one-on-one sessions, the health educator empower patients to pre-empt situations that have been shown to lead to non-adherence and make plans for situations in which they are less likely to adhere.

Components of the E-ASP

The E-ASP augments S-ASP and consistS of several interconnected components: 1) development and maintenance of an educational and supportive milieu at the CDC Clinic, 2) provision of five structured education, support and behavioural skills building sessions, and (3) three weekly ART planning sessions.

Development and Maintenance of an Educational and Supportive Milieu

A separate room is available for exclusive use of the E-ASP. This room has educational materials available at all times, and is a comfortable area for patients to relax and socialize with one another during the course of their time at the CDC clinic.

Provision by Study Health Educator of 5 Structured Education, Support, and Behavioural Skills Sessions

The educational, support, and behavioural skills building sessions consist of five, one-on-one interactive sessions that will be conducted by the health educator. The sessions take place at five important times during patients' early ART:

1. On the day of commencement of ART - "Preparing to take ART medications"
2. 2 weeks after starting ART - "Adjusting to taking ART medications"
3. 2 months after starting ART - "Feeling good and staying healthy taking ART medications"
4. 3 months after starting ART - "Planning for ongoing HIV care and daily ART medications"
5. 6 months after starting ART - "Preparation for lifelong HIV care and daily ART medications"

The content matter (key educational, support and skills points/messages) for the sessions is conveyed by the study health educator using specially designed story board flip charts, put into table-standing easel display books; the front side faces the patient and the backside faces the health educator. Posters including all pertinent images and messages will be put onto the walls for ease of summarizing the information, and for providing an overview of important messages. All messages will also be conveyed in pictorial form to ensure that literacy levels of the cohort do not negatively affect understanding.

The other important educational, motivation and skills building tool available is a double-sided Adherence Problem Solving Pocket Card. This tool lists commonly occurring medication adherence problems on the front side and practical solutions/strategies on the back.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the CAPRISA CAT programme and the CDC.
* Willing and able to provide written consent to take part in the study.
* > 18 years of age (to give consent for participation)
* Eligible for initiation of HAART (currently CD4+ <200)

Exclusion Criteria:

* Unwillingness or inability to adhere to the study schedule

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 297 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
suppressed viral load at 9 months | 9 months
  Those participants with suppressed viral load at 9 months will be classed as treatment success, all others will be classed as treatment failures for the purposes of this outcome.

SECONDARY OUTCOMES:
feasibility of E-ASP in this resource constrained setting | one year
Secondly to describe the relationship between adherence and viral load and CD4+counts | 2 months, 9 months and 12 months
describe factors associated with poor/good adherence in this group | one year
describe the relationship between early adherence and adherence at subsequent timepoints | 2 weeks, and 2 and 9 months after start ART and 12 months
to establish the validity of self-reported adherence (in relation to pill counts) in this context | one year
to assess the long-term impact of E-ASP on adherence | 18 months
suppressed viral load at 12 months | 12 months
  Those participants with suppressed viral load will be classed at treatment successes, all others will be classed as treatment failures for this secondary outcome measure.
adherence at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francois van Loggerenberg, MA(ResPsych), Principal Investigator — CAPRISA, University of KwaZulu-Natal
Locations (1):
- CAPRISA eThekwini Clinical Research Site, Durban, KwaZulu-Natal, South Africa

REFERENCES:
- [Background] Amico KR, Toro-Alfonso J, Fisher JD. An empirical test of the information, motivation and behavioral skills model of antiretroviral therapy adherence. AIDS Care. 2005 Aug;17(6):661-73. doi: 10.1080/09540120500038058. PMID 16036253
- [Result] van Loggerenberg F, Grant AD, Naidoo K, Murrman M, Gengiah S, Gengiah TN, Fielding K, Abdool Karim SS. Individualised motivational counselling to enhance adherence to antiretroviral therapy is not superior to didactic counselling in South African patients: findings of the CAPRISA 058 randomised controlled trial. AIDS Behav. 2015 Jan;19(1):145-56. doi: 10.1007/s10461-014-0763-6. PMID 24696226
- See also: Primary outcome paper — http://link.springer.com/article/10.1007/s10461-014-0763-6